CLINICAL TRIAL: NCT06728553
Title: A Pilot, Phase 2a, Randomized, Double-blind, Placebo-controlled, Cross-over Clinical Study to Evaluate Safety and Efficacy of Sublingual MTX101 for the Acute Treatment of Migraine Headaches in Adults
Brief Title: Safety and Efficacy Trial of MTX101 2mg for the Acute Treatment of Migraine in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Manistee Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MTX101-0202 / Pro00082158
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Migraine
Keywords: acute treatment of migraine; nervous system diseases; central nervous system diseases; brain diseases; headache; migraine with or without aura
MeSH Terms: conditions — Migraine Disorders; Nervous System Diseases; Central Nervous System Diseases; Brain Diseases; Headache

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects will be given one sublingual tablet of matching placebo and instructed to take the tablet after the onset of a migraine of moderate to severe intensity.
  Interventions: Drug: Placebo
- Active (Experimental): Subjects will be given one 2 mg sublingual tablet of the investigational product (MTX101) and instructed to take the tablet after onset of a migraine of moderate to severe intensity.
  Interventions: Drug: MTX101

INTERVENTIONS:
Drug: MTX101 — One 2 mg sublingual tablet of MTX101
  Arms: Active
Drug: Placebo — One sublingual tablet of placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if drug MTX101 works to treat acute migraine attacks in adults. It will also learn about the safety of the drug MTX101. The main questions it aims to answer are:

Does the drug MTX101 lower headache pain for participants and the need to use a rescue medication? What side effects, if any, do participants have when taking the drug MTX101? Researchers will compare the drug MTX101 to a placebo (a look-alike substance that contains no drug) to see if the drug MTX101 works to treat acute migraine attacks.

Participants will:

Take the drug MTX101 or a placebo to treat 1 migraine attack with each treatment.

Visit the clinic twice and have one phone call over a 4 week period for checkups and tests.

Keep a diary of their symptoms and the number of times they use a rescue medication.

DETAILED DESCRIPTION:
Subjects enrolled in the study will be randomized to receive investigational product (MTX101 2mg or placebo), to be taken as soon as they have a migraine headache that reaches moderate to severe intensity. Subjects will take a single dose of either active or placebo to treat one migraine headache. Rescue medication should not be taken until at least 2 hours post study medication dose.

The subject will have a telephone check up within 72 to 120 hours after treatment of the first migraine headache.

The subject will treat a 2nd moderate to severe migraine at least 48 hours after the first treated migraine headache.

The subject will return to the clinic for re-evaluation within a 4 week period from the start of the study.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female aged 18 to 65 years at the time of consent.
2. Onset of migraine headache before age 50.
3. History of episodic migraine headache starting at least 1-year ago with or without aura.
4. Has a minimum of 4 monthly migraine days and not more than 10 migraine days per month.
5. Able to distinguish pain related to migraine attacks from tension-type and cluster headache attacks.
6. Able to understand and provide signed informed consent.
7. Willing and able to comply with all scheduled visits, treatment plan, and other study procedures.

Key Exclusion Criteria:

1. No more than a total of 15 headache days per month.
2. Use of more than 2 migraine preventive medications.
3. Current diagnosis of glaucoma.
4. Use of opioids or barbiturates more than 4 days/month, triptans or ergots 10 or more days/month, or simple analgesics (e.g., aspirin, NSAIDs, acetaminophen) 15 or more days/month in the 3 months prior to Visit 1.
5. Current diagnosis of any post-traumatic headaches, medication overuse headaches, new daily persistent headache, trigeminal autonomic cephalgia (e.g., cluster headache), painful cranial neuropathy or daily headaches.
6. Vaccination within less than 7 days from the Screening or plans to get a vaccine during the study or within a week after final study dose.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Safety assessment (occurrence of adverse events, treatment emergent adverse events and serious adverse events). | Treatment emergent adverse event safety assessments will be limited to the first 48 hours after a treated attack.
  To assess the tolerability and safety of MTX101. This objective will be measured by assessing the number of unique subjects with deaths, serious adverse events, and moderate and severe adverse events.

SECONDARY OUTCOMES:
The change in migraine headache pain score, using an 11-point Numerical Rating Scale, (0=no pain, 10=worst possible pain). | From the time of dosing (t=0 hour) to 2 hours post-dose.
  This objective will be measured by change in migraine headache pain score, using an 11-point Numerical Rating Scale, (0=no pain, 10=worst possible pain), from the time of dosing (t=0 hour) to 2 hours post-dose as recorded on the subject's Diary.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Sponsor GmbH
Locations (7):
- United States (7):
  - Kaizen Brain Center, La Jolla, California
  - Clinical Research Institute, LLC, Santa Monica, California
  - Brainstorm Research, Miami, Florida
  - Synergy Clinical Research/Emerald Coast Center for Neurological Disorders, Pensacola, Florida
  - DelRicht Research, New Orleans, Louisiana
  - QUEST Research Institute, Farmington Hills, Michigan
  - Wasatch Clinical Research, Salt Lake City, Utah